CLINICAL TRIAL: NCT00426764
Title: A Phase II, Multicenter, Open-Label Trial Evaluating The Activity And Tolerability Of Romidepsin (Depsipeptide, FK228) In Progressive Or Relapsed Peripheral T-Cell Lymphoma Following Prior Systemic Therapy (GPI-06-0002)
Brief Title: A Trial of Romidepsin for Progressive or Relapsed Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPI-06-0002; 2006-006228-21 (EudraCT Number); NCT00924378 (obsolete NCT alias)
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: peripheral T-cell lymphoma; T-cell lymphoma; romidepsin
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — romidepsin; Depsipeptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Romidepsin (Experimental): Participants received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — Romidepsin intravenously (through a vein) over 4 hours on Days 1, 8 and 15 of each 28-day cycle.
  Other Names: ISTODAX; Depsipeptide; FK228

SUMMARY:
The purpose of this study is to evaluate the activity of romidepsin in patients with progressive or relapsed peripheral T-cell lymphoma (PTCL) who have already been treated with systemic therapy.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, open-label, single-arm trial. This study is designed on the basis of complete response (CR) or unconfirmed CR [CR(u)] as the measure of efficacy, based on the best overall response of each patient. The sample size of 65 patients evaluable for efficacy would yield lower 95% confidence limits on the rate of CR + CR(u) that would range from 2.2% to 7.7%, if the observed rate of CR + CR(u) ranges from 8% to 15%. The study was amended to include an Extension Phase, during which patients at non-US sites who are benefitting from treatment can continue to receive romidepsin. The Extension Study Phase is active in EU countries where currently no Marketing Authorisation exists for romidepsin. Patients may remain on study until progressive disease occurs or they withdraw their consent and only serious adverse events and study drug administration data will continue to be collected and reported for these patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for study participation and have:

* Histologically confirmed PTCL not otherwise specified, angioimmunoblastic T-cell lymphoma, extranodal natural killer (NK)/T-cell lymphoma nasal type, enteropathy- type T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, cutaneous γδ T-cell lymphoma (excludes mycosis fungoides or Sezary syndrome), transformed mycosis fungoides, hepatosplenic T-cell lymphoma, anaplastic large cell lymphoma (ALCL; anaplastic lymphoma kinase [ALK]-1 negative), or patients with ALK 1 expressing ALCL (ALK-1 positive) who have relapsed disease after autologous stem cell transplant (ASCT);
* Age ≥18 years;
* Written informed consent;
* Progressive disease following at least one systemic therapy or refractory to at least one prior systemic therapy;
* Measurable disease according to the International Workshop Response (IWC) criteria and/or measurable cutaneous disease;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Serum potassium ≥3.8 mmol/L and magnesium ≥0.85 mmol/L (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria);
* Negative urine or serum pregnancy test on females of childbearing potential; and
* All women of childbearing potential must use an effective barrier method of contraception (either an intrauterine contraceptive device [IUCD] or double barrier method using condoms or a diaphragm plus spermicide) during the treatment period and for at least 1 month thereafter. Male patients should use a barrier method of contraception during the treatment period and for at least 1 month thereafter. Hormonal methods of contraception such as the contraceptive pill or patch (particularly those containing ethinyl-estradiol) should be avoided due to a potential drug interaction.

Exclusion Criteria:

Patients are ineligible for entry if any of the following criteria are met:

* Known central nervous system (CNS) lymphoma [computed tomography (CT) or magnetic resonance imaging (MRI) scans are required only if brain metastasis is suspected clinically];
* Chemotherapy or immunotherapy within 4 weeks of study entry (6 weeks if nitrosoureas given);
* Initiation of corticosteroids during study (defined as 7 days prior to Cycle 1 Day 1[C1D1] until study drug discontinuation)

  * Patients treated with a pulse of steroids were to discontinue steroid use 7 days prior to C1D1 and have a repeat CT scan and disease assessment after discontinuation of corticosteroids and before starting romidepsin;
* Concomitant use of any other anti-cancer therapy;
* Concomitant use of any investigational agent;
* Use of any investigational agent within 4 weeks of study entry;
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome;
  * QTc interval >480 milliseconds (msec);
  * A myocardial infarction within 6 months of C1D1. Patients with a history of myocardial infraction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate;
  * Other significant electrocardiogram (ECG) abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
  * Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV. In any patient in whom there is doubt, the patient should be referred to a cardiologist for evaluation;
  * An ECG recorded at screening showing significant ST depression (ST depression of ≥2 mm, measured from isoelectric line to the ST segment at a point 60 msec at the end of the QRS complex). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI;
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  * Hypertrophic cardiomyopathy or restrictive cardiomyopathy from prior treatment or other causes (if in doubt, see ejection fraction criteria above);
  * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria;
  * Any cardiac arrhythmia requiring anti-arrhythmic medication;
* Serum potassium <3.8 mmol/L or serum magnesium <0.85 mmol/L (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria);
* Concomitant use of drugs that may cause a significant prolongation of the QTc;
* Concomitant use of CYP3A4 significant or moderate inhibitors;
* Concomitant use of therapeutic warfarin or another anticoagulant due to a potential drug interaction. Use of a small dose of a anticoagulant to maintain patency of venous access port and cannulas is permitted;
* Clinically significant active infection;
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C;
* Previous extensive radiotherapy involving ≥30% of bone marrow (e.g., whole pelvis, half spine), excluding patients who have had total body irradiation as part of a conditioning regimen for ASCT;
* Major surgery within 2 weeks of study entry;
* Previous allogeneic stem cell transplant;
* Inadequate bone marrow or other organ function as evidenced by:

  * Hemoglobin <9 g/dL (transfusions and/or erythropoietin are permitted);
  * Absolute neutrophil count (ANC) ≤1.0 × 10^9 cells/L [patients with neutropenia (ANC 1-1.5 10^9 cells/L) as a function of their disease may be supported with granulocyte-colony stimulating factor (G-CSF)];
  * Platelet count <100 × 10^9 cells/L or platelet count <75 × 10^9 cells/L if bone marrow disease involvement is documented;
  * Total bilirubin >2.0 × upper limit of normal (ULN) or >3.0 × ULN in the presence of demonstrable liver metastases;
  * Aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) >2.0 × ULN or >3.0 × ULN in the presence of demonstrable liver metastases; or
  * Serum creatinine >2.0 × ULN;
* Patients who are pregnant or breast-feeding;
* Coexistent second malignancy or history of prior solid organ malignancy within previous 3 years (excluding basal or squamous cell carcinoma of the skin, and in situ carcinoma of the cervix (CIN 1) that has been treated curatively);
* Any prior history of a hematologic malignancy (other than T-cell lymphoma);
* Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures; or
* Prior exposure to romidepsin (other histone deacetylase inhibitors are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-06-19 (Actual); Primary Completion 2010-11-11 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Czuczman, MD, Study Director — Celgene
Locations (90):
- United States (45):
  - Moore UCSD Cancer Center, La Jolla, California
  - UCLA Division of Hematology Oncology, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University IRB, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cancer Centers of Florida, PA, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta Oncology Associates, P.C., Augusta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Cancer Care and Hematology Specialists of Chicagoland, Arlington Heights, Illinois
  - Hematology Oncology Assoc. of IL Orchard Research LLC, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - St. Agnes - Medical Center, Baltimore, Maryland
  - Center for Cancer And Blood Disorders, Bethesda, Maryland
  - Center for Cancer Research CAMC, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, PA, Burnsville, Minnesota
  - St. Joseph Oncology, Inc, Saint Joseph, Missouri
  - Arch Medical Services, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Taussig Cancer Center Cleveland Clinic Foundation, Cleveland, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Accelerated Community Oncology Research Network Inc ACORN, Memphis, Tennessee
  - Mamie McFadden Ward Center, Beaumont, Texas
  - Methodist Charlton Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center Simmons Comprehensive Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology, P.A.-Fort Worth, Fort Worth, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - Allison Cancer Center, Midland, Texas
  - US Oncology, Plano, Texas
  - HOAST, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology, PA, Waco, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (4):
  - Mater Private Medical Centre - Haematology and Oncology Clinics of Australasia Research Centre, South Brisbane, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne
  - St. Vincent Hospital, Fitzroy
  - Royal North Shore Hospital, St Leonards
- Czechia (4):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital of Kralovske Vinohrady, Prague
  - Charles University General Hospital, Prague
- France (9):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - CHU Nantes Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Service des Maladies du Sang, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
- Germany (7):
  - Charite Universitatsmedizin Berlin campus Virchow Klinikum Centrum fur Tumormedizin, Berlin
  - Uniklinik Koln, Cologne
  - Krankenhaus Nordwest, Frankfurt a.M.
  - Georg-August-Universität Göttingen, Göttingen
  - Klinikum der Universitat Munchen-Grosshadern, München
  - Klinikum Nurnberg Nord, Nuremberg
  - UKT Universitaetsklinikum Tuebingen, Tübingen
- Poland (4):
  - Klinika Hematologii Akademickie Centrum Kliniczne Akademii Medycznej w Gdansku, Gdansk
  - Oddzial Kliniczny Kliniki Hematologii, Krakow
  - Wojewodzki Szpital Specjalistczny im. Mikolaja Kopernika, Lodz
  - Klinika Nowotworow Ukladu Chlonnego, Warsaw
- Spain (6):
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santandar
- Sweden (2):
  - Lund University Hosptial, Lund
  - Akademiska Sjukhuset, Uppsala
- Ukraine (4):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - National Cancer Institute Department Of Conservative Methods Of Treatment, Kyiv
  - R.E.Kavetsky Institute of Experimental Pathology, Oncology and Radiobiology, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine of the AMS of Ukraine, Lviv
- United Kingdom (5):
  - Barts Cancer Institute, Queen Mary University of London, Charterhouse Square, London
  - Guy's and St. Thomas' Hospital, London
  - Catherine Lewis Centre - Hematology Department, London
  - Royal Free Hospital, London Hampstead
  - Somers Cancer Research Building, Southampton

REFERENCES:
- [Background] Foss F, Pro B, Miles Prince H, Sokol L, Caballero D, Horwitz S, Coiffier B. Responses to romidepsin by line of therapy in patients with relapsed or refractory peripheral T-cell lymphoma. Cancer Med. 2017 Jan;6(1):36-44. doi: 10.1002/cam4.939. Epub 2016 Dec 16. PMID 27981793
- [Background] Shustov A, Coiffier B, Horwitz S, Sokol L, Pro B, Wolfson J, Balser B, Eisch R, Popplewell L, Prince HM, Allen SL, Piekarz R, Bates S. Romidepsin is effective and well tolerated in older patients with peripheral T-cell lymphoma: analysis of two phase II trials. Leuk Lymphoma. 2017 Oct;58(10):2335-2341. doi: 10.1080/10428194.2017.1295143. Epub 2017 Mar 7. PMID 28264616
- [Result] Coiffier B, Pro B, Prince HM, Foss F, Sokol L, Greenwood M, Caballero D, Borchmann P, Morschhauser F, Wilhelm M, Pinter-Brown L, Padmanabhan S, Shustov A, Nichols J, Carroll S, Balser J, Balser B, Horwitz S. Results from a pivotal, open-label, phase II study of romidepsin in relapsed or refractory peripheral T-cell lymphoma after prior systemic therapy. J Clin Oncol. 2012 Feb 20;30(6):631-6. doi: 10.1200/JCO.2011.37.4223. Epub 2012 Jan 23. PMID 22271479
- [Result] Horwitz S, Coiffier B, Foss F, Prince HM, Sokol L, Greenwood M, Caballero D, Morschhauser F, Pinter-Brown L, Iyer SP, Shustov A, Nichols J, Balser J, Balser B, Pro B. Utility of (1)(8)fluoro-deoxyglucose positron emission tomography for prognosis and response assessments in a phase 2 study of romidepsin in patients with relapsed or refractory peripheral T-cell lymphoma. Ann Oncol. 2015 Apr;26(4):774-779. doi: 10.1093/annonc/mdv010. Epub 2015 Jan 20. PMID 25605745
- [Derived] Foss F, Horwitz S, Pro B, Prince HM, Sokol L, Balser B, Wolfson J, Coiffier B. Romidepsin for the treatment of relapsed/refractory peripheral T cell lymphoma: prolonged stable disease provides clinical benefits for patients in the pivotal trial. J Hematol Oncol. 2016 Mar 10;9:22. doi: 10.1186/s13045-016-0243-8. PMID 26965915
- [Derived] Foss F, Coiffier B, Horwitz S, Pro B, Prince HM, Sokol L, Greenwood M, Lerner A, Caballero D, Baran E, Kim E, Nichols J, Balser B, Wolfson J, Whittaker S. Tolerability to romidepsin in patients with relapsed/refractory T-cell lymphoma. Biomark Res. 2014 Sep 8;2:16. doi: 10.1186/2050-7771-2-16. eCollection 2014. PMID 25279222
- [Derived] Coiffier B, Pro B, Prince HM, Foss F, Sokol L, Greenwood M, Caballero D, Morschhauser F, Wilhelm M, Pinter-Brown L, Padmanabhan Iyer S, Shustov A, Nielsen T, Nichols J, Wolfson J, Balser B, Horwitz S. Romidepsin for the treatment of relapsed/refractory peripheral T-cell lymphoma: pivotal study update demonstrates durable responses. J Hematol Oncol. 2014 Jan 23;7:11. doi: 10.1186/1756-8722-7-11. PMID 24456586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Romidepsin
Started | 131 (Represents the number of patients who received any amount of study drug.)
Discontinued Prior to or During Cycle 6 | 98
Discontinued at End of or After Cycle 6 | 33
Completed | 0
Not Completed | 131
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 6
Not completed — Compassionate Use | 1
Not completed — Progressive Disease | 83
Not completed — Adverse Event | 24
Not completed — Other | 1
Not completed — Death | 1
Not completed — Other Reasons (Miscellaneous) | 10

BASELINE CHARACTERISTICS:
Groups:
- Romidepsin: Participants received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Participants who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
Arm/Group | Romidepsin
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 116
  Black | 7
  Asian | 3
  Other | 4
  Unknown | 1
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: participants with a Baseline measurement
  m^2
    number analyzed (Participants) | 128
    (all) | 1.84 (0.2348)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — The ECOG scale is as follows: Grade 0: Fully active, able to carry on all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or Chair.
  Participants
    0 | 46
    1 | 66
    2 | 17
    Missing | 1
    Unknown | 1
Duration of peripheral T-cell lymphoma (PTCL) [Mean (Standard Deviation); unit: years] | 2.268 (2.6654)
PTCL Subtype Based on Central Diagnosis [Count of Participants; unit: Participants] — ALK-1=anaplastic lymphoma kinase; ALCL=anaplastic large cell lymphoma
  Participants
    PTCL Unspecified (NOS) | 69
    Angioimmunoblastic T-cell lymphoma (AITL) | 27
    ALK-1 negative ALCL | 21
    Enteropathy-type T-cell lymphoma | 6
    Subcutaneous panniculitis-like T-cell lymphoma | 3
    ALK-1 positive ALCL | 1
    Cutaneous γδ T-cell lymphoma | 1
    Extranodal NK/T cell lymphoma nasal type | 1
    Transformed mycosis fungoides | 1
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response According to the International Workshop Response Criteria (IWC) for Non-Hodgkin's Lymphomas (NHL) Assessed by an Independent Review Committee
Description: Complete Response (CR): >75% decrease in size aggregate of nodal index lesions (large and small), complete disappearance of extranodal and non-index lesions; total disappearance of clinical disease including skin involvement; disease-related signs and symptoms, normalization of biochemical abnormalities and reduction in size of spleen or liver so no longer palpable. Unconfirmed CR: all above criteria except all nodal index lesions must have regressed >75% in the sum of the product diameters (SPD) from baseline. Individual nodes previously confluent must have regressed by >75% in their SPD.
Time Frame: Response was assessed after every 2 cycles of treatment and at completion of therapy, up until 30 September 2012 (data cutoff for analysis). Maximum duration on study was 1931 days.
Population: Histologically Confirmed Population, comprised all enrolled patients who received at least 1 dose of study treatment and who had histopathologically confirmed peripheral T-cell lymphoma(s). Patients who discontinued prior to any response evaluation or who had no post-baseline assessment of response were classified as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 130
percentage of participants | 15.4 [9.7 to 22.8]

2. Secondary Outcome: Percentage of Participants With Objective Disease Response
Description: Objective disease response was defined as patients with a Complete Response, Unconfirmed Complete Response or a Partial Response (PR) according to the IWC 1999 assessed by an independent review committee: CR, Cru defined above, PR defined as ≥50% decrease in size of 6 largest dominant nodes and/or nodal masses & extranodal index lesions and no increase of non-index lesions, liver, or spleen; no new sites of disease evident; skin lesions decreased by ≥50%.
Time Frame: as for outcome 1
Population: Histologically Confirmed Population. Patients who discontinued prior to any response evaluation or who had no post-baseline assessment of response were classified as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 130
percentage of participants | 26.2 [18.8 to 34.6]

3. Secondary Outcome: Duration of Objective Disease Response
Description: Duration of response was defined as the number of days from the date of the first disease response (Complete, Unconfirmed Complete or Partial Response) until the date of progression and was determined using Kaplan-Meier product-limit estimates. Progression was defined as: a ≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions.
Time Frame: as for outcome 1
Population: Histopathologically-Confirmed Population with an objective response. Censoring for patients who did not have a date of progression was conducted based on last assessment reported for the patient.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Romidepsin
Number analyzed (Participants) | 34
days | NA [353 to NA] — The median and the upper limit of the 95% confidence interval were not estimable due to the low number of events.

4. Secondary Outcome: Duration of Complete Disease Response
Description: Duration of response was defined as the number of days from the date of the first disease response (Complete or Unconfirmed Complete) until the date of progression and was determined using Kaplan-Meier product-limit estimates. Progression was defined as: a ≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions.
Time Frame: as for outcome 1
Population: Histopathologically-Confirmed Population with a complete response. Censoring for patients who did not have a date of progression was conducted based on last assessment reported for the patient.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Romidepsin
Number analyzed (Participants) | 20
days | NA [500 to NA] — Median and upper limit of the 95% confidence interval was not estimable due to the low number of events.

5. Secondary Outcome: Time to Disease Progression
Description: Time to progression (≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions) was defined as the duration from the date of the first study drug dose to the date of relapse or progression as reported by the independent review committee and was determined using Kaplan-Meier product-limit estimates.
Time Frame: as for outcome 1
Population: Histopathologically-Confirmed Population. Censoring for patients who did not have a date of progression was conducted based on last assessment reported for the patient.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Romidepsin
Number analyzed (Participants) | 130
days | 182 [106 to 290]

6. Secondary Outcome: Change in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG scale is as follows: Grade 0: Fully active, able to perform all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory, able to carry out light work; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair. Data reported is the shift from Baseline ECOG score to best on-study assessment score.
Time Frame: From Baseline up until 30 September 2012 (data cutoff for analysis). Maximum duration on study was 1931 days.
Population: Safety Population: all participants who received at least 1 dose of romidepsin.
Measure: Number; unit: participants
Groups:
- Missing: Participants with a missing best on study ECOG performance score, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
- Best ECOG = 0: Participants with a best on study ECOG performance score of 0, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
- Best ECOG = 1: Participants with a best on study ECOG performance score of 1, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
- Best ECOG = 2: Participants with a best on study ECOG performance score of 2, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
- Best ECOG = 3: Participants with a best on study ECOG performance score of 3, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
- Best ECOG = 4: Participants with a best on study ECOG performance score of 4, who received romidepsin 14 mg/m^2 administered intravenously over 4 hours on Days 1, 8, and 15 of a 28-day cycle. Participants continued on monthly cycles of romidepsin. The planned duration of study therapy was 6 cycles. Patients who responded could continue beyond 6 cycles until disease progression or other withdrawal criteria were met. For participants treated for 12 or more cycles, maintenance dosing (2 doses per cycle) was permitted.
Arm/Group | Missing | Best ECOG = 0 | Best ECOG = 1 | Best ECOG = 2 | Best ECOG = 3 | Best ECOG = 4
Number analyzed (Participants) | 5 | 40 | 57 | 19 | 6 | 4
participants
  Missing Baseline ECOG Score | 1 | 0 | 0 | 0 | 0 | 0
  Baseline ECOG Score = 0 | 2 | 26 | 16 | 1 | 0 | 1
  Baseline ECOG Score = 1 | 1 | 13 | 35 | 12 | 4 | 2
  Baseline ECOG Score = 2 | 1 | 1 | 6 | 6 | 2 | 1
  Baseline ECOG Score = 3 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline ECOG Score = 4 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event or experience (AE) is defined as any untoward medical occurrence, which does not necessarily have to have a causal relationship with this treatment. A serious AE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event or condition. Related AEs are defined as those considered by the Investigator to have a possible, probable, or very likely/certain relationship to the study drug. AEs were graded as mild (1), moderate (2), severe (3), lifethreatening (4), or death (5). TEAEs occurred from the first dose of study medication through the end of the study (30 days post last dose) or any event that was present at baseline but worsened in intensity or was subsequently considered drug-related by the Investigator through end of study.
Time Frame: From first dose of study treatment until the final study visit, which occurred 30 days after receiving the last dose. Mean duration of treatment up until 30 September 2012 (data cutoff for analysis) was 169 days.
Population: Safety Population: all participants who received at least 1 dose of romidepsin.
Measure: Count of Participants; unit: Participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 131
Participants
  TEAE | 128
  ≥ Grade 3 TEAE | 89
  ≥ Grade 4 TEAE | 27
  Serious TEAE | 61
  TEAE Leading to Discontinuation | 25
  Deaths within 30 days of Last Dose | 8

ADVERSE EVENTS:
Time Frame: Adverse events were reported and documented throughout the study from first dose of study treatment until the final study visit, which occurred 30 days after receiving the last dose. The mean duration of treatment was 210 days.
Description: NOTE: events shown include data from 6 participants who were ongoing in study treatment at the time of the last data cut-off (30-Sep-2012), which updated the mean duration of treatment from 196 to 210 days.
Arm/Group | Romidepsin
All-Cause Mortality (participants affected / at risk) | 9/131
Serious Adverse Events (participants affected / at risk) | 62/131
Other Adverse Events (participants affected / at risk) | 124/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin (N=131)
Anaemia (Blood and lymphatic system disorders) | 3
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Subendocardial ischaemia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 1
Chest pain (General disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 11
Cytokine release syndrome (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Candida sepsis (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 5
Erysipelas (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 6
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Aspiration tracheal (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Electrocardiogram repolarisation abnormality (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Magnesium deficiency (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Deep vein thrombosis (Vascular disorders) | 5
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin (N=131)
Anaemia (Blood and lymphatic system disorders) | 32
Leukopenia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 53
Tachycardia (Cardiac disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 15
Abdominal pain upper (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 39
Diarrhoea (Gastrointestinal disorders) | 46
Dyspepsia (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 76
Stomatitis (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 48
Asthenia (General disorders) | 22
Chest pain (General disorders) | 8
Chills (General disorders) | 14
Fatigue (General disorders) | 53
Oedema (General disorders) | 7
Oedema peripheral (General disorders) | 13
Pain (General disorders) | 10
Pyrexia (General disorders) | 44
Nasopharyngitis (Infections and infestations) | 7
Oral candidiasis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 7
Weight decreased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 38
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 27
Headache (Nervous system disorders) | 19
Lethargy (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Skin lesion (Skin and subcutaneous tissue disorders) | 11
Hypotension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation.